CLINICAL TRIAL: NCT02990169
Title: Clinical Evaluation of CATS Tonometer Prism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CATS and Corneal Thickness
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Ocular Hypotension
MeSH Terms: conditions — Ocular Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Goldmann Tonometer (Active Comparator): determine if the CATS tonometer prism effectively reduces sensitivity to IOP errors produced by corneal thickness and therefore provides a more accurate IOP reading compared to the reference tonometer (Goldmann prism), based upon the correction value table for Goldmann tonometer prism
  Interventions: Device: Goldmann Tonometer prism
- CATS tonometer (Active Comparator): determine if the CATS tonometer prism effectively reduces sensitivity to IOP errors produced by corneal thickness and therefore provides a more accurate IOP reading compared to the reference tonometer (Goldmann prism), based upon the correction value table for Goldmann tonometer prism
  Interventions: Device: CATS tonometer prism

INTERVENTIONS:
Device: CATS tonometer prism — IOP tonometer prism for assessment of intraocular pressure
  Arms: CATS tonometer
Device: Goldmann Tonometer prism — IOP tonometer prism for assessment of intraocular pressure
  Arms: Goldmann Tonometer

SUMMARY:
Prospective, open-labeled, randomized, controlled, multicenter study at two clinical investigative sites in Tucson, Arizona. The subjects will undergo intraocular pressure measurement with the CATS tonometer prism and the Goldmann applanation tonometer prism (GAT). Seventy-five (75) Subjects 18 and older and will be enrolled. Subjects will be screened based on standard of care vision examination at the clinical investigation sites. All subjects will undergo a standard ophthalmic exam and informed consent. IOP will be measured using a Goldmann tonometer armature with both the standard flat GAT prism and the modified curved CATS prism alternately inserted. The only additional measurement is central corneal thickness (CCT) which is used to correct for one of the corneal biomechanical errors seen in the GAT prism and is currently standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Male and female patients, at least 18 years of age

Exclusion Criteria:

* Subject has undergone ocular surgery within the last 3 months
* Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's heath at risk
* Pregnant or nursing women
* Subjects with only one functional eye
* Those with one eye having poor or eccentric fixation
* Eyes displaying an oval contact image
* Those with corneal scarring or who have had corneal surgery including corneal laser surgery
* Microphthalmos
* Buphthalmos
* Contact lens wearers
* Severe Dry eyes
* Lid squeezers - blepharospasm
* Nystagmus
* Keratoconus
* Any other corneal or conjunctival pathology or infection.
* Central corneal thickness between 0.600 mm and 0.500 mm (more than 2 standard deviations about the human mean)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
All subjects will have CATS tonometer prism intraocular pressure readings compared to Goldmann tonometer prism readings. | From date of randomization until 24 hours
All subjects will have corneal thickness measurements performed and the CATS tonometer prism intraocular pressure readings will be compared to Goldmann tonometer readings using a correction value table. | From date of randomization until 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Eye Consultants, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCafferty SJ, Tetrault K, McColgin A, Chue W, Levine J, Muller M. Modified Goldmann prism intraocular pressure measurement accuracy and correlation to corneal biomechanical metrics: multicentre randomised clinical trial. Br J Ophthalmol. 2019 Dec;103(12):1840-1844. doi: 10.1136/bjophthalmol-2018-313470. Epub 2019 Feb 22. PMID 30796054